CLINICAL TRIAL: NCT03706430
Title: Validation of RPVi as a Parameter to Predict Fluid Responsiveness
Status: Terminated | Type: Interventional
Why Stopped: Sponsor requested
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CANN0011
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Surgery; Anesthesia

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Pulse Co-Oximeter sensor (Experimental): All subjects are enrolled into this arm and will receive an investigational pulse CO-Oximeter sensors.
  Interventions: Device: Pulse CO-Oximeter sensor

INTERVENTIONS:
Device: Pulse CO-Oximeter sensor — Investigational Pulse CO-Oximeter sensor will measure hemoglobin (SpHb), Pulse Rate (PR), Perfusion Index (Pi), Methemoglobin (SpMet), Pleth Variability Index (PVi), RPVi, etc.

SUMMARY:
This is a prospective, nonrandomized, sequential data collection study to evaluate the ability of RPVi to predict fluid responsiveness in comparison with other dynamic parameters including stroke volume variation (SVV) and/or pulse pressure variation (PPV).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of consent
* Scheduled for elective surgery requiring general anesthesia and mechanical ventilation
* Arterial line and other standard of care line placement indicated as part of the scheduled surgical procedure

Exclusion Criteria:

* Patients diagnosed with or history of heart failure, angina, pulmonary heart disease, rheumatic heart disease, cardiomyopathy, congenital heart disease, or valvular heart disease.
* Patients scheduled for or has had a liver transplant
* Patients with surgeries at or around site of sensor placement or skin abnormalities affecting the sensor placement area such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails that would prevent monitoring of pulse-oximeter physiological parameters during the study.
* Patients with cardiac arrhythmias
* Patients with intracardiac shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulse Co-Oximeter Sensor
Started | 63
Completed | 48
Not Completed | 15
Not completed — No A-Line placed | 5
Not completed — Subject had gel nail polish | 1
Not completed — Nail length causing difficulties with sensor | 1
Not completed — Cancelled Case | 6
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pulse Co-Oximeter Sensor
Number analyzed (Participants) | 48
Age, Customized [Count of Participants; unit: Participants]
  ≤ 18 years | 0
  Between 18 and 65 years | 23
  ≥ 65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of RPVi to SVV and/or PPV
Description: To evaluate the ability of RPVi to predict fluid responsiveness in comparison with other dynamic parameters including Stroke Volume Variation (SVV) and/or Pulse Pressure Variation (PPV) using Bland Altman analysis.
Time Frame: approximately 2-6 hours during surgery
Population: Zero subjects were collected for validation as the study was terminated in the data collection phase due to slow enrollment
Arm/Group | Pulse Co-Oximeter Sensor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2-6 hours during surgery
Arm/Group | Pulse Co-Oximeter Sensor
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03706430/Prot_SAP_000.pdf